CLINICAL TRIAL: NCT05486663
Title: The Effect of the Tactile/kinesthetic Stimulus Program on the Maturation of Sucking Ability in Preterm Infants
Brief Title: Tactile/kinesthetic Stimulus Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gonca Karatas Baran (Other)
Responsible Party: Sponsor-Investigator, Gonca Karatas Baran, Dr Nurse, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEONATAL CARE
Record Dates: First submitted 2022-07-29; First posted 2022-08-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Breast Feeding, Exclusive; Enteral Feeding; Hospital Stay
Keywords: breasfeeding; enteral feeding; tactile/kinesthetic intervention
MeSH Terms: conditions — Breast Feeding | interventions — Touch

STUDY DESIGN:
Intervention Model Description: There will be two group. One is intervential group, other is control group
Who Masked: Participant
Masking Description: The volunteer (newborn's mother or father) will not know which group she/he will be in before joining the study. After accepting to the participate in the study, the volunteer will be informed abouth which group her/his newborn will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tactile/kinesthetic Group (Experimental): After the stability of the general health status of the babies is ensured and the oral feeding decision is made, tactile / kinesthetic application will be made for 14 days, 2 times a day, for 15 minutes just before feeding.
  Interventions: Other: Tactile/kinesthetic Group
- Control Group (No Intervention): Tactile / kinesthetic applications will not be applied to the control group and these babies will be followed for 14 days and at discharge after the stability of the general health status of the babies is ensured and the oral feeding decision is made.

INTERVENTIONS:
Other: Tactile/kinesthetic Group — Tactile/kinesthetic stimulation is performed in three stages. In the first stage; for tactile stimulation; The baby is placed in the prone (prone) position in the incubator. Light massage was applied in the head, shoulder, back, legs and arms of the infants. Each massage is applied 12 times for 1 minute. Massage was performed for 5 seconds. In the second stage Kinesthetic stimulation, including elbow flexion-extension movement, palm massages, flexion-extension of the knees and legs and plantar massages, was applied while the neonate was in supine position. Each kinesthetic stimulation was performed for 5 seconds. Each movement was repeated six times, with a total duration of 5 minutes. Tactile stimulation was repeated once after kinesthetic stimulation. The total duration of TKS was 15 minutes which was performed three times daily preferably between breastfeeding or bottle feeding for 14 consecutive days.
  Other Names: Case
  Arms: Tactile/kinesthetic Group

SUMMARY:
The study will be carried out as a prospective randomized controlled clinical study to determine the effect of tactile/kinesthetic stimulus program on preterm infants on transition time to full sucking, sucking success and hospital stay.

DETAILED DESCRIPTION:
Application of the Research Tactile/kinesthetic Group After the stability in the general health status of the babies and the oral feeding decision are made, for 14 days, 2 times a day, just before feeding; There will be a 15-minute tactile/kinesthetic application. Complications that may develop during the tactile/kinesthetic application in infants will be monitored by evaluating the physical findings of the preterm infant and on the bedside monitor. In cases such as decreased oxygen saturation, apnea and bradycardia during the tactile/kinesthetic intervention, the procedure will not be performed or will be delayed until the baby regains stability.

Note: The application will be carried out by showing the necessary sensitivity for the preterm baby (not shaking the baby, not moving the baby suddenly, the temperature of the hands being close to the baby's body temperature, etc.) and by the researcher nurses experienced in NICU.

Control Group Tactile/kinesthetic applications will not be applied to the control group and these babies will be followed up for 14 days and at discharge after the stability of the general health status of the babies is ensured and the oral feeding decision is made.

In both groups; Baby scales and tape measure will be used for anthropometric measurement of body weight before and after breastfeeding. Other data will be obtained from the patient file and observations made during the hospitalization of the preterm infant.

The LATCH Breastfeeding Diagnosis Form (during the first mother's breastfeeding) will be filled in by observation, by the researcher and an observer nurse, as it is an observation-based form. The researcher will train the observer on the use of the LATCH Breastfeeding Diagnostic Form. The researcher and observer will simultaneously and independently evaluate each preterm infant by scoring the LATCH Breastfeeding Diagnostic Form during the breastfeeding period. In order to evaluate the agreement among the observers, the agreement will be evaluated by looking at Cohen's Kappa coefficient. The LATCH second measurement will be made on Day 5.

The amount of food taken during breastfeeding within 14 days (1st, 5th, 9th, 13th, and on the day of discharge) will be determined by measuring body weight before and after feeding. Body weight will be weighed before and after feeding at discharge. The times of full enteral feeding and full oral feeding will be recorded in the groups.

Hypotheses H0 hypothesis: Tactile/kinesthetic stimulus interventions have no effect on transition time to full oral feeding in preterm infants.

Hypothesis H1: In preterm infants, interventions with tactile/kinesthetic stimuli have an effect on transition time to full oral feeding.

ELIGIBILITY:
Inclusion criteria

* Born between 28-32 weeks of gestation,
* Stable vital signs,
* 1st and 5th minute APGAR score between 6-10,
* Babies who have received mechanical ventilator or continuous positive air pressure (CPAP) or both support after 48 hours have passed after stabilization,
* Does not have an anomaly that will prevent feeding,
* Oral feeding decision has been made,
* Babies of mothers who are willing to breastfeed their babies,
* Babies of parents who volunteered to participate in the study will be taken.

Exclusion criteria

* IUGG,
* Infants with severe asphyxia,
* Babies born with low birth weight according to their gestational week,
* Having an anomaly that will prevent her from feeding,
* Babies with unstable vital signs,
* Babies with congenital anomalies or serious complications
* Infants with intraventricular bleeding.

Dismissal Criteria

• Babies whose oral feeding process is interrupted for more than 1 day due to neonatal problems.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
transition time (day) to full oral feeding | within the first 30 days of birth
  This is the data on which day full oral feeding is started after admission to the neonatal intensive care unit.
transition time(day) to oral feeding trials | within the first 30 days of birth
  This is the data on which day oral feeding trials were performed after admission to the neonatal intensive care unit. intensive care unit.
transition time (day) to full enteral feeding | within the first 30 days of birth
  This is the data on which day full enteral feeding is started after admission to the neonatal intensive care unit.
transition time (day) to enteral feeding trials | within the first 30 days of birth
  This is the data on which day full enteral feeding is started after admission to the neonatal intensive care unit.
time (day) to first breastfeeding | within the first 30 days of birth
  This is the data on which day breastfeeding feeding is started after admission to the neonatal intensive care unit.
latch score (first day of breastfeeding) | first breastfeeding process (20 minutes)
  Using LATCH Scale. The minimum LATCH score is 0 and the maximum is 10.
latch score (fifth day of breastfeeding) | fifth day breastfeeding process (20 minutes)
  Using LATCH Scale. The minimum LATCH score is 0 and the maximum is 10.
length of hospital stay (days) | the date of at discharge (up to 40 weeks)
  length of hospital stay (days)
change in weight before and after feeding | the date of at discharge (up to 40 weeks)
  babies will be weighed before and after feeding on the first, fifth, ninth, thirteenth day and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: GONCA K KARATAS BARAN, Study Director — Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Locations (1):
- Etlık Zubeyde Hanım Kadın Hastalıkları Eğitim Ve Araştırma Hastanesi, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bond C. Positive Touch and massage in the neonatal unit: a British approach. Semin Neonatol. 2002 Dec;7(6):477-86. doi: 10.1053/siny.2002.0149. PMID 12614600
- [Background] Burklow KA, McGrath AM, Kaul A. Management and prevention of feeding problems in young children with prematurity and very low birth weight. Inf Young Children. 2002; 14(4):19-30.
- [Background] Clark GF, Avery-Smith W, Wolf LS, Anthony P, Holm SE, Hertfelder SD, Youngstrom MJ; Eating and Feeding Task Force; Commission on Practice. Specialized knowledge and skills in eating and feeding for occupational therapy practice. Am J Occup Ther. 2003 Nov-Dec;57(6):660-78. doi: 10.5014/ajot.57.6.660. No abstract available. PMID 14661785
- [Background] Diego MA, Field T, Hernandez-Reif M. Vagal activity, gastric motility, and weight gain in massaged preterm neonates. J Pediatr. 2005 Jul;147(1):50-5. doi: 10.1016/j.jpeds.2005.02.023. PMID 16027695
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Fuccile S. Pre-feeding Sensorimotor Stimulation as an Early Intervention Strategy to Enhance Oral Feeding Skills in Preterm Infants. Health Sciences - Occupational Health and Therapy, doctoral thesis, McGill University, QC, Canada, 2008
- [Background] Gewolb IH, Vice FL. Abnormalities in the coordination of respiration and swallow in preterm infants with bronchopulmonary dysplasia. Dev Med Child Neurol. 2006 Jul;48(7):595-9. doi: 10.1017/S0012162206001241. PMID 16780630
- [Background] Jaywant SS, Kale JS.The effect of pre-feeding protocol with andwithout tactile and kinaesthetic stimulation onoral motor ability & physiological stability inpreterm infants. Int J Health Sci Res. 2021;11(1):38-4
- [Background] Mathai S, Fernandez A, Mondkar J, Kanbur W. Effects of tactilekinesthetic stimulation in preterms: a controlled trial. Indian Pediatr. 2001; 38(10),:1091-1098. • McGrath JM, Braescu AV. State of the science: feeding readiness in the preterm infant. J Perinat Neonatal Nur. 2004;18(4):353-368
- [Background] Bache M, Pizon E, Jacobs J, Vaillant M, Lecomte A. Effects of pre-feeding oral stimulation on oral feeding in preterm infants: a randomized clinical trial. Early Hum Dev. 2014 Mar;90(3):125-9. doi: 10.1016/j.earlhumdev.2013.12.011. Epub 2014 Jan 23. PMID 24461572